CLINICAL TRIAL: NCT02926586
Title: Fludarabine and Cytarabine Versus High-dose Cytarabine in Consolidation Treatment of Core-bing Factor Acute Myeloid Leukemia: A Prospective, Multicenter, Randomized Study
Brief Title: Fludarabine and Cytarabine Versus High-dose Cytarabine for CBF-AML
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBF-AML-2016
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia; Core-Binding Factor
Keywords: RUNX1-RUNX1T1; CBFβ-MYH11; fludarabine; cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; fludarabine phosphate; Cytarabine

ARMS (2):
- Fludarabine (Experimental): The patients in experimental arm should receive the consolidation chemotherapy regimen with fludarabine and cytarabine. The dosage of fludarabine is 30mg/m2/d for 5 days intravenously and cytarabine is 1500mg/m2/d for 5 days intravenously.
  Interventions: Drug: Fludarabine
- high-dose cytarabine (Active Comparator): The patients in control arm should receive the consolidation chemotherapy regimen with high-dose cytarabine. The dosage of cytarabine is 2000mg/m2/12h for 3 days (1,3,5) intravenously.
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 50 mg/m2, IV (in the vein) in combination with cytarabine 1500mg/m2/d for 5 days with each cycle of 28 days. Number of cycles: 4
  Other Names: Fludara
  Arms: Fludarabine
Drug: Cytarabine — 2000mg/m2/12h, IV (in the vein) for 3 days with each cycle of 28 days. Number of cycles: 4
  Other Names: Cytosar
  Arms: high-dose cytarabine

SUMMARY:
The purpose of the study is to determine whether Fludarabine in combination with cytarabine is more effective than high-dose cytarabine in post-remission therapy for patients with core-binding factor acute myeloid leukemia

DETAILED DESCRIPTION:
The recurrence rate, relapse-free survival rate, and overall survival rate of CBF-AML patients were compared between FA and HIDAC regimens. Observe the prognostic value of factors such as c-KIT gene mutation and minimal residual disease (MRD).

ELIGIBILITY:
Inclusion Criteria:

* Clinical and laboratory diagnosis of CBF-AML,including RUNX1-RUNX1T1 and CBF-MYH11 fusion gene rearrangement by PCR/FISH
* In status of complete remission after one to two courses of induction therapy
* Total bilirubinic acid ≤ 35μmol/L, AST/ALT<2 times abnormal level, serum creatinine < 1.5mg/ml
* Cardiac function: EF ≥ 50%
* Hydroxyurea can be used for patient with white blood cell count ≥ 50*109/L
* ECOG (Eastern Cooperative Oncology Group) score: ≤ 2

Exclusion Criteria:

* Relapsed/refractory AML
* Serious liver/ kidney dysfunction
* Cardiac function level: 2 above
* Female in pregnancy or lactation
* With serious infection diseases or other diseases
* Not obey the principle of clinical study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with disease recurrence | one year
  Comparing the percentage of participants with disease recurrence with two therapeutic regimen

SECONDARY OUTCOMES:
Percentage of Participants in survival | one year
  Comparing the percentage of Participants in survival with two therapeutic regimen

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, Doctor, Principal Investigator — Department of hematology, Shanghai General Hospital, No. 100 Haining Road, Shang
Locations (1):
- Xianmin Song, Shanghai, Shanghai Municipality, China